CLINICAL TRIAL: NCT01042691
Title: A Phase I Trial of Isolated Hepatic Perfusion With Oxaliplatin Followed by Hepatic Arterial Infusion of FUDR and Leucovorin for Patients With Unresectable Colorectal Liver Metastases
Brief Title: Isolated Liver Perfusion With Oxaliplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: David Bartlett (Other)
Collaborators: The Pittsburgh Foundation (Other); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, David Bartlett, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-135
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Unresectable Colorectal Liver Metastases
MeSH Terms: interventions — Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxaliplatin (Experimental): Subjects who are planning to undergo surgery for placement of HAI therapy pump will be considered for enrollment. Standard HAI therapy requires a laparotomy and placement of an intrahepatic arterial catheter that is connected to one of several commercially available subcutaneous electronic pumps. The pump is then used to deliver FUDR and Leucovorin directly to the liver, usually beginning four weeks after surgery and lasts on average for a period of six to twelve months after the study. This study will examine the addition of a one hour isolated hepatic perfusion with oxaliplatin to this standard treatment
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — The starting dose of oxaliplatin administered via isolated hepatic perfusion will be the safe tolerated dose of intra-arterial infusion and pharmacokinetics from intravenous studies. The dose will be 5 mg/m2 and will be escalated.

SUMMARY:
The primary goal of this research study is to determine a safe dose for the drug oxaliplatin when delivered by isolated hepatic perfusion. The second goal of this research study is to determine if isolated hepatic perfusion with oxaliplatin can improve the efficacy of standard hepatic arterial infusional (HAI) therapy with floxuridine (FUDR)/leucovorin.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included that are scheduled to undergo surgery for placement of hepatic arterial infusion pump for HAI therapy and
* Histologically or cytologically proven measurable metastatic colorectal cancer limited to the parenchyma of the liver with no evidence of unresectable extrahepatic disease by preoperative radiological studies. Limited resectable extrahepatic disease is acceptable.
* No chemotherapy, radiotherapy, or biologic therapy for their malignancy in the 4 weeks prior to the liver perfusion and must have recovered from all side effects.
* An ECOG performance standard of 0, 1 or 2 for 24 hours prior to surgery.
* Adequate hepatic function as evidenced by bilirubin < 2.0 mg/dL and a PT < 2 seconds greater than the upper limit of normal.
* Age equal to 18 years or older and greater than 30 kg.
* Platelet counts greater than 100,000, a hematocrit > 27.0, a white blood count > 3000/microliter, and a creatinine less than or equal to 1.5 mg/dL or a creatinine clearance of > 60 mL/min. Patients with elevations in hepatic transaminases secondary to the presence of metastatic disease in the liver are eligible.
* Aware of the neoplastic nature of his/her illness, the experimental nature of the therapy, alternative treatments, potential benefits, and risks and willing to sign an informed consent.
* The disease in the liver must be considered unresectable as defined by greater than three sites of disease in the liver, bilobar disease, and tumor abutting major vascular or ductal structures making anatomic resection with preservation of liver function impossible.

Exclusion Criteria:

* Pregnant patients and nursing mothers will be excluded due to the unknown effects of oxaliplatin on the fetus or newborn
* Patients taking immunosuppressive drugs or on chronic anticoagulation will not be eligible.
* Patients with active infections are not eligible.
* Patients with biopsy proven cirrhosis or evidence of significant portal hypertension manifested by ascites, esophageal varices on endoscopy, or radiologic studies showing significant collateral vessels around the organs drained by the portal venous system will be excluded.
* Patients with ischemic cardiac disease or history of congestive heart failure with an LVEF < 40% will be excluded.
* Patients with COPD or other chronic pulmonary disease with PFT's indicating an FEV< 50% predicted for age will be excluded.
* Patients with a history of veno-occlusive disease of the liver are ineligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and dose limiting toxicity of oxaliplatin delivered via isolated hepatic perfusion (IHP). | 12 months

SECONDARY OUTCOMES:
To determine if isolated hepatic perfusion with oxaliplatin can increase the response rate, duration of response and survival of patients being treated with standard HAI with FUDR when compared to historical controls. | 2-3 years
To determine the tissue absorption of oxaliplatin in normal liver versus tumor during IHP. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David L Bartlett, M.D., Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Lahr CJ, Soong SJ, Cloud G, Smith JW, Urist MM, Balch CM. A multifactorial analysis of prognostic factors in patients with liver metastases from colorectal carcinoma. J Clin Oncol. 1983 Nov;1(11):720-6. doi: 10.1200/JCO.1983.1.11.720. PMID 6668490
- [Background] Blumgart LH, Fong Y. Surgical options in the treatment of hepatic metastasis from colorectal cancer. Curr Probl Surg. 1995 May;32(5):333-421. doi: 10.1016/s0011-3840(05)80012-7. PMID 7538062
- [Background] Choti MA, Bulkley GB. Management of hepatic metastases. Liver Transpl Surg. 1999 Jan;5(1):65-80. doi: 10.1002/lt.500050113. PMID 9873095
- [Background] Bartlett DL. Treatment of patients with hepatic metastases. Cancer J. 2000 Apr;6 Suppl 2:S169-76. No abstract available. PMID 10803832
- [Background] Balch CM, Urist MM, Soong SJ, McGregor M. A prospective phase II clinical trial of continuous FUDR regional chemotherapy for colorectal metastases to the liver using a totally implantable drug infusion pump. Ann Surg. 1983 Nov;198(5):567-73. doi: 10.1097/00000658-198311000-00001. PMID 6227295
- [Background] Kemeny,M.M., S.Adak, and S.Lipsitz. 1999. Results of the intergroup [Eastern Cooperative Oncology Group (ECOG) and Southwest Oncology Group (SWOG) prospective randomized study of surgery alone versus continuous hepatic artery infusion of FuDR and continuous systemic infusion of 5FU after hepatic resection for colorectal liver metastases. Proc ASCO 18:1012.
- [Background] Lokich JJ, Sonneborn H, Paul S, Zipoli T. Phase I study of continuous venous infusion of floxuridine (5-FUDR) chemotherapy. Cancer Treat Rep. 1983 Sep;67(9):791-3. PMID 6224555
- [Background] Alexander HR Jr, Fraker DL, Bartlett DL. Isolated limb perfusion for malignant melanoma. Semin Surg Oncol. 1996 Nov-Dec;12(6):416-28. doi: 10.1002/(SICI)1098-2388(199611/12)12:63.0.CO;2-D. PMID 8914206
- [Background] Alexander HR Jr, Bartlett DL, Libutti SK, Fraker DL, Moser T, Rosenberg SA. Isolated hepatic perfusion with tumor necrosis factor and melphalan for unresectable cancers confined to the liver. J Clin Oncol. 1998 Apr;16(4):1479-89. doi: 10.1200/JCO.1998.16.4.1479. PMID 9552055
- [Background] Bartlett DL, Libutti SK, Figg WD, Fraker DL, Alexander HR. Isolated hepatic perfusion for unresectable hepatic metastases from colorectal cancer. Surgery. 2001 Feb;129(2):176-87. doi: 10.1067/msy.2001.110365. PMID 11174711
- [Background] Raymond E, Chaney SG, Taamma A, Cvitkovic E. Oxaliplatin: a review of preclinical and clinical studies. Ann Oncol. 1998 Oct;9(10):1053-71. doi: 10.1023/a:1008213732429. PMID 9834817
- [Background] Rixe O, Ortuzar W, Alvarez M, Parker R, Reed E, Paull K, Fojo T. Oxaliplatin, tetraplatin, cisplatin, and carboplatin: spectrum of activity in drug-resistant cell lines and in the cell lines of the National Cancer Institute's Anticancer Drug Screen panel. Biochem Pharmacol. 1996 Dec 24;52(12):1855-65. doi: 10.1016/s0006-2952(97)81490-6. PMID 8951344
- [Background] Kern W, Beckert B, Lang N, Stemmler J, Beykirch M, Stein J, Goecke E, Waggershauser T, Braess J, Schalhorn A, Hiddemann W. Phase I and pharmacokinetic study of hepatic arterial infusion with oxaliplatin in combination with folinic acid and 5-fluorouracil in patients with hepatic metastases from colorectal cancer. Ann Oncol. 2001 May;12(5):599-603. doi: 10.1023/a:1011186708754. PMID 11432616
- [Background] Rietbroek RC, van de Vaart PJ, Haveman J, Blommaert FA, Geerdink A, Bakker PJ, Veenhof CH. Hyperthermia enhances the cytotoxicity and platinum-DNA adduct formation of lobaplatin and oxaliplatin in cultured SW 1573 cells. J Cancer Res Clin Oncol. 1997;123(1):6-12. doi: 10.1007/BF01212608. PMID 8996534
- [Background] Urano M, Ling CC. Thermal enhancement of melphalan and oxaliplatin cytotoxicity in vitro. Int J Hyperthermia. 2002 Jul-Aug;18(4):307-15. doi: 10.1080/02656730210123534. PMID 12079586
- [Background] Elias D, Bonnay M, Puizillou JM, Antoun S, Demirdjian S, El OA, Pignon JP, Drouard-Troalen L, Ouellet JF, Ducreux M. Heated intra-operative intraperitoneal oxaliplatin after complete resection of peritoneal carcinomatosis: pharmacokinetics and tissue distribution. Ann Oncol. 2002 Feb;13(2):267-72. doi: 10.1093/annonc/mdf019. PMID 11886004
- [Background] Alexander,H.R., D.L.Bartlett, D.L.Fraker, S.K.Libutti, T.Moser, and S.A.Rosenberg. 1997. Results of a Phase II study of isolated hepatic perfusion (IHP) with tumor necrosis factor (TNF) and melphalan for unresectable primary or metastatic cancer confined to the liver. Proc.Soc.Surg.Oncol. 6:8. (Abstr.)
- [Background] Alexander HR, Libutti SK, Bartlett DL, Puhlmann M, Fraker DL, Bachenheimer LC. A phase I-II study of isolated hepatic perfusion using melphalan with or without tumor necrosis factor for patients with ocular melanoma metastatic to liver. Clin Cancer Res. 2000 Aug;6(8):3062-70. PMID 10955785
- [Background] Erkmen K, Egorin MJ, Reyno LM, Morgan R Jr, Doroshow JH. Effects of storage on the binding of carboplatin to plasma proteins. Cancer Chemother Pharmacol. 1995;35(3):254-6. doi: 10.1007/BF00686557. PMID 7805185